CLINICAL TRIAL: NCT06871072
Title: Telerehabilitation for Multiple Sclerosis: Artificial Intelligence vs. Conventional Approaches in Strength Training. A Sin-gle-Blinded Randomized Clinical Trial
Brief Title: Telerehabilitation for Multiple Sclerosis
Acronym: TRHBN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: v.1 -11/12/2023
Record Dates: First submitted 2025-02-27; First posted 2025-03-11 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
Keywords: artificial intelligence; exercise; multiple sclerosis; physical therapy; strength; telerehabilitation
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Telerehabilitation; Resistance Training

STUDY DESIGN:
Intervention Model Description: A neurology will be diagnosed the Multiple sclerosis .
Masking Description: Enter the total number of arms participants might be assigned to over the course of the clinical study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (Experimental): EG performed using an artificial intelli-gence (AI) application called RehBody, which detects body segments, assists in cor-recting the technique and monitoring the exercise, number of sets and repetitions done, and the adherence percentage.
  Interventions: Other: Telerehabilitation
- Control group (Active Comparator): CG participants followed the exercise program and trained at home with images and videos as support.
  Interventions: Other: Exercise program

INTERVENTIONS:
Other: Telerehabilitation — EG performed using an artificial intelli-gence (AI) application called RehBody, which detects body segments, assists in cor-recting the technique and monitoring the exercise, number of sets and repetitions done, and the adherence percentage
  Arms: Telerehabilitation
Other: Exercise program — CG participants followed the exercise program and trained at home with images and videos as support.
  Arms: Control group

SUMMARY:
Multiple sclerosis (MS) is a neurodegenerative disease affecting the central nervous system and is a leading cause of disability in young adults. It often produces strength deficits. Exercise has been shown to improve strength, mobility, and quality of life while reducing fatigue. Telerehabilitation offers a convenient, accessible alternative for MS patients. This study explores the use of an AI-powered application for prescribing and monitoring strength exercises, ensuring continuous feedback and adherence. Methods: Randomized clinical trial. Intervention of 3 weekly strength training ses-sions for 20 weeks, patients in the experimental group used the AI application, while patients in the control group followed the conventional method, paper-based exercises with access to videos.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis according to the McDonald criteria 2017:
* Age between 35 and 60 years.
* Score on the Expanded Disability Status Scale in Multiple Sclerosis by Kurtzke (EDSS) between 2 and 6 points.
* Patients who do not require assistive devices for home mobility.
* Patients with no changes in disease-modifying treatment in the last 3 months.
* Patients who have understood, completed, and signed the informed consent and the study information sheet.

Exclusion Criteria:

* Patients who have been regularly performing strength exercises for more than 3 months prior.
* Moderate/severe cognitive impairment that may interfere with the understanding and/or execution of the study.
* History of alcohol and/or drug abuse.
* Presence of a relapse and/or treatment with corticosteroids within the four weeks prior to the start of the study.
* Patients with severe comorbidities other than MS that may pose a risk for following the exercise guidelines or for their participation in the study for other reasons.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 58 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Maximal Strength | Baseline
  Maxi-mal Strength was assessed using an 8-repetition maximum test , in which par-ticipants perform 8 repetitions of squat and bench press as the resistance is gradually increased until a load is determined where only eight repetitions can be performed. The load increment was determined based on the result from the Modified Borg Scale at the end of the exercise, if the Borg rating was greater than 7, the test was completed.

SECONDARY OUTCOMES:
Maximal Strength. | Ten weeks.
  Maxi-mal Strength was assessed using an 8-repetition maximum test, in which par-ticipants perform 8 repetitions of squat and bench press as the resistance is gradually increased until a load is determined where only eight repetitions can be performed. The load increment was determined based on the result from the Modified Borg Scale at the end of the exercise, if the Borg rating was greater than 7, the test was completed.
Maximal Strength. | Twenty weeks.
  Maxi-mal Strength was assessed using an 8-repetition maximum test, in which par-ticipants perform 8 repetitions of squat and bench press as the resistance is gradually increased until a load is determined where only eight repetitions can be performed. The load increment was determined based on the result from the Modified Borg Scale at the end of the exercise, if the Borg rating was greater than 7, the test was completed.
Strength endurance. | Baseline
  Strength endurance was measured by the maximum number of unilateral knee flexion-extension repetitions performed in 30 seconds
Endurance capacity. | Baseline.
  Endurance capacity as secondary variable was measured by 6-minutes walking test , where participants covering the maximum distance on a flat surface in 6 minutes. Fatigue was quantified by Modified Fatigue Impact Scale .
Strength endurance. | ten weeks
  Strength endurance was measured by the maximum number of unilateral knee flexion-extension repetitions performed in 30 seconds
Strength endurance. | twenty weeks.
  Strength endurance was measured by the maximum number of unilateral knee flexion-extension repetitions performed in 30 seconds
Endurance capacity. | ten weeks
  Endurance capacity as secondary variable was measured by 6-minutes walking test , where participants covering the maximum distance on a flat surface in 6 minutes. Fatigue was quantified by Modified Fatigue Impact Scale.
Endurance capacity. | Twenty weeks
  Endurance capacity as secondary variable was measured by 6-minutes walking test, where participants covering the maximum distance on a flat surface in 6 minutes. Fatigue was quantified by Modified Fatigue Impact Scale

CONTACTS AND LOCATIONS:
Overall Officials: Lucía Ortega Carrión, Physiotherapy, Principal Investigator — Hospital Universitario macarena del servicio Andaluz de Salud
Locations (1):
- Macarena University Hospital, Seville, Spain

REFERENCES:
- [Background] Compston A, Coles A. Multiple sclerosis. Lancet. 2008 Oct 25;372(9648):1502-17. doi: 10.1016/S0140-6736(08)61620-7. PMID 18970977
- [Background] Dilokthornsakul P, Valuck RJ, Nair KV, Corboy JR, Allen RR, Campbell JD. Multiple sclerosis prevalence in the United States commercially insured population. Neurology. 2016 Mar 15;86(11):1014-21. doi: 10.1212/WNL.0000000000002469. Epub 2016 Feb 17. PMID 26888980
- [Background] Meier S, Willemse EAJ, Schaedelin S, Oechtering J, Lorscheider J, Melie-Garcia L, Cagol A, Barakovic M, Galbusera R, Subramaniam S, Barro C, Abdelhak A, Thebault S, Achtnichts L, Lalive P, Muller S, Pot C, Salmen A, Disanto G, Zecca C, D'Souza M, Orleth A, Khalil M, Buchmann A, Du Pasquier R, Yaldizli O, Derfuss T, Berger K, Hermesdorf M, Wiendl H, Piehl F, Battaglini M, Fischer U, Kappos L, Gobbi C, Granziera C, Bridel C, Leppert D, Maleska Maceski A, Benkert P, Kuhle J. Serum Glial Fibrillary Acidic Protein Compared With Neurofilament Light Chain as a Biomarker for Disease Progression in Multiple Sclerosis. JAMA Neurol. 2023 Mar 1;80(3):287-297. doi: 10.1001/jamaneurol.2022.5250. PMID 36745446
- [Background] Rodriguez Murua S, Farez MF, Quintana FJ. The Immune Response in Multiple Sclerosis. Annu Rev Pathol. 2022 Jan 24;17:121-139. doi: 10.1146/annurev-pathol-052920-040318. Epub 2021 Oct 4. PMID 34606377
- [Background] Thompson AJ, Banwell BL, Barkhof F, Carroll WM, Coetzee T, Comi G, Correale J, Fazekas F, Filippi M, Freedman MS, Fujihara K, Galetta SL, Hartung HP, Kappos L, Lublin FD, Marrie RA, Miller AE, Miller DH, Montalban X, Mowry EM, Sorensen PS, Tintore M, Traboulsee AL, Trojano M, Uitdehaag BMJ, Vukusic S, Waubant E, Weinshenker BG, Reingold SC, Cohen JA. Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria. Lancet Neurol. 2018 Feb;17(2):162-173. doi: 10.1016/S1474-4422(17)30470-2. Epub 2017 Dec 21. PMID 29275977
- [Background] Lublin FD, Reingold SC, Cohen JA, Cutter GR, Sorensen PS, Thompson AJ, Wolinsky JS, Balcer LJ, Banwell B, Barkhof F, Bebo B Jr, Calabresi PA, Clanet M, Comi G, Fox RJ, Freedman MS, Goodman AD, Inglese M, Kappos L, Kieseier BC, Lincoln JA, Lubetzki C, Miller AE, Montalban X, O'Connor PW, Petkau J, Pozzilli C, Rudick RA, Sormani MP, Stuve O, Waubant E, Polman CH. Defining the clinical course of multiple sclerosis: the 2013 revisions. Neurology. 2014 Jul 15;83(3):278-86. doi: 10.1212/WNL.0000000000000560. Epub 2014 May 28. PMID 24871874
- [Background] Podbielska M, O'Keeffe J, Pokryszko-Dragan A. New Insights into Multiple Sclerosis Mechanisms: Lipids on the Track to Control Inflammation and Neurodegeneration. Int J Mol Sci. 2021 Jul 7;22(14):7319. doi: 10.3390/ijms22147319. PMID 34298940
- [Background] Boissy AR, Cohen JA. Multiple sclerosis symptom management. Expert Rev Neurother. 2007 Sep;7(9):1213-22. doi: 10.1586/14737175.7.9.1213. PMID 17868019
- [Background] Galea I, Ward-Abel N, Heesen C. Relapse in multiple sclerosis. BMJ. 2015 Apr 14;350:h1765. doi: 10.1136/bmj.h1765. No abstract available. PMID 25872511
- [Background] Lizak N, Lugaresi A, Alroughani R, Lechner-Scott J, Slee M, Havrdova E, Horakova D, Trojano M, Izquierdo G, Duquette P, Girard M, Prat A, Grammond P, Hupperts R, Grand'Maison F, Sola P, Pucci E, Bergamaschi R, Oreja-Guevara C, Van Pesch V, Ramo C, Spitaleri D, Iuliano G, Boz C, Granella F, Olascoaga J, Verheul F, Rozsa C, Cristiano E, Flechter S, Hodgkinson S, Amato MP, Deri N, Jokubaitis V, Spelman T, Butzkueven H, Kalincik T; MSBase Study Group. Highly active immunomodulatory therapy ameliorates accumulation of disability in moderately advanced and advanced multiple sclerosis. J Neurol Neurosurg Psychiatry. 2017 Mar;88(3):196-203. doi: 10.1136/jnnp-2016-313976. Epub 2016 Sep 28. PMID 27683916
- [Background] Halabchi F, Alizadeh Z, Sahraian MA, Abolhasani M. Exercise prescription for patients with multiple sclerosis; potential benefits and practical recommendations. BMC Neurol. 2017 Sep 16;17(1):185. doi: 10.1186/s12883-017-0960-9. PMID 28915856